CLINICAL TRIAL: NCT03263637
Title: A Phase 1, Open-Label, Multicentre, Non-Randomized Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of AZD4573, a Potent and Selective CDK9 Inhibitor, in Subjects With Relapsed or Refractory Haematological Malignancies
Brief Title: Study to Assess Safety, Tolerability, Pharmacokinetics and Antitumor Activity of AZD4573 in Relapsed/Refractory Haematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8230C00001
Record Dates: First submitted 2017-08-11; First posted 2017-08-28 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Relapsed or Refractory Haematological Malignancies Including; Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; High Risk Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Richter's Syndrome; B-cell Non-Hodgkin Lymphoma; T-cell Non-Hodgkin Lymphoma; Small Lymphocytic Lymphoma; Multiple Myeloma
Keywords: Relapsed or refractory haematological malignancies; AZD4573; CDK9i; Acute Myeloid Leukemia (AML); Acute Lymphocytic Leukemia (ALL); Chronic lymphocytic Leukemia (CLL); High risk Myelodysplastic syndrome (MDS); Chronic Myelomonocytic Leukemia (CML); Richter's syndrome; B-cell Non-Hodgkin Lymphoma (B-cell NHL); T-cell Non-Hodgkin Lymphoma (T-cell NHL); Small lymphocytic Lymphoma (SLL); Multiple Myeloma (MM)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelomonocytic, Chronic; Lymphoma, B-Cell; Lymphoma, T-Cell; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This study is a multicentre, open-label, first in human, non-randomized, dose-escalation study including an intra-subject ramp-up. The study will consist of two, parallel dose escalation arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: (Cohort 1-3) (Experimental): dose level 1-3 in subjects with relapsed or refractory haematological malignancies excluding AML/ALL/high-risk MDS/CMML/CLL.
  Interventions: Drug: AZD4573
- Arm B: (Cohort 1-3) (Experimental): dose level 1-3 in subjects with relapsed or refractory AML, ALL, high-risk MDS, CMML, CLL and Richter's syndrome.
  Interventions: Drug: AZD4573

INTERVENTIONS:
Drug: AZD4573 — AZD4573 will be administered as a intravenous (IV) infusion.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary antitumor activity of AZD4573 in subjects with relapsed or refractory haematological malignancies.

ELIGIBILITY:
Main Inclusion Criteria (cohorts 1, 2, 3):

• Patients with histologically confirmed, relapsed or refractory haematological malignancies. Patients will include but are not limited to the following: Arm A : B-cell Non-Hodgkin lymphoma , T-cell Non-Hodgkin lymphoma , Small lymphocytic lymphoma (SLL) , Multiple myeloma (MM) Arm B: CLL (chronic lymphocytic leukaemia), Richter's syndrome , AML/secondary AML, ALL , High-risk myelodysplastic syndrome (MDS), CMML (chronic myelomonocytic leukemia)

* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Must have received at least 2 prior lines of therapy
* Documented active disease requiring treatment per respective NCCN/ESMO guideline that is relapsed or refractory defined as: Recurrence of disease after response to prior line(s) of therapy Or progressive disease after completion of the treatment regimen preceding entry into the study
* Adequate hematologic, hepatic and renal function
* Women should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test before start of dosing if of child-bearing potential or must have evidence of nonchildbearing potential
* Men should be willing to use barrier contraception (ie, condoms) and refrain from sperm donation during and after the conduct of the trial.

Main Exclusion Criteria (cohorts 1,2, 3):

* Treatment with any of the following: any other chemotherapy, immunotherapy or anticancer agents within 2 weeks, any hematopoietic growth factors (e.g., filgrastim; [G-CSF] or sargramostin [GM-CSF]) within 7 days of the first dose of investigational product or pegylated G-CSF (pegfilgrastim) or darbepoetin within 14 days, any full-dose level anti-coagulation treatment sufficiently prior to treatment that INR is <1.5 (DVT/PE prophylaxis dose is allowed) or Major surgery (excluding placement of vascular access) within 4 weeks (with regard to the first dose of study treatment on this protocol).
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment.
* Presence of, or history of, CNS lymphoma, leptomeningeal disease or spinal cord compression.
* History of prior nonhematologic malignancy with exceptions mentioned in protocol
* Undergone any procedures or experienced any of the conditions listed in protocol exclusion criteria currently or in the preceding 6 months
* Patients with any of the following: evidence of severe or uncontrolled systemic disease, asecretory myeloma, a known history of infection with human immunodeficiency virus (HIV), serological evidence of active Hepatitis B infection, cardiac abnormalities as mentioned in the protocol, previous allogeneic bone marrow transplant, adrenal gland insufficiency or pancreatitis.
* History of severe allergic or anaphylactic reactions to BH3 mimetics or history of hypersensitivity to active or inactive excipients of AZD4573.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | At every treatment and follow up visit from the time of informed consent up to 8 months initially or if clinical benefit continues, until disease progression. Expected to be for 12 months
  Number of subjects with adverse events as a measure of safety and tolerability including changes in vital signs, electrocardiograms (ECGs), safety and laboratory parameters
Dose limiting toxicities | From day 1 of first cycle for a period of 8 weeks for cohorts 1 and 2, and for a period of 4 weeks for cohort 3 and for any other subsequent cohort that may be opened
  DLTs will be determined from monitoring adverse events (AEs), and abnormal laboratory tests (clinical chemistry, hematology, and urinalysis), physical examinations, vital signs (blood pressure and pulse), and electrocardiogram (ECG).
Maximum tolerated dose | After completion of dose limiting toxicity (DLT) period (8/4 weeks) for the maximum dose cohort

SECONDARY OUTCOMES:
Maximum observed plasma concentration of AZD4573 | For Cohorts 1 and 2: Over 8 weeks (from dosing Day 1 of ramp-up Cycle A until Day 1 of the target dose Cycle 1). For Cohort 3: Over 4 weeks (from dosing Day 1 of ramp-up Cycle A until Day 1 of the target dose Cycle 1)
  The concentration of AZD4573 and its metabolites in blood will be determined (Cmax will be derived).
Area under the concentration-time curve for plasma concentrations of AZD4573 | For Cohorts 1 and 2: Over 8 weeks (from dosing Day 1 of ramp-up Cycle A until Day 1 of the target dose Cycle 1). For Cohort 3: Over 4 weeks (from dosing Day 1 of ramp-up Cycle A until Day 1 of the target dose Cycle 1).
  The Area under the curve of AZD4573 and its metabolites in blood will be determined
Volume of distribution (Vd). | For Cohorts 1 and 2: Over 8 weeks (from dosing Day 1 of ramp-up Cycle A until Day 1 of the target dose Cycle 1). For Cohort 3: Over 4 weeks (from dosing Day 1 of ramp-up Cycle A until Day 1 of the target dose Cycle 1).
  The concentration of AZD4573 and its metabolites in blood will be determined. Volume of distribution (Vd) is the apparent volume in which a drug is distributed (i.e., the parameter relating drug concentration to drug amount in the body).
Clearance (CL). | For Cohorts 1 and 2: Over 8 weeks (from dosing Day 1 of ramp-up Cycle A until Day 1 of the target dose Cycle 1). For Cohort 3: Over 4 weeks (from dosing Day 1 of ramp-up Cycle A until Day 1 of the target dose Cycle 1).
  The concentration of AZD4573 and its co-former in blood will be determined. Clearance (CL) is the volume of plasma cleared of the drug per unit time.
Antitumor activity of AZD4573 in patients by assessing overall response rate (ORR). | From time of first dose until discontinuation of AZD4573 expected to be for up to 12 months
  To assess proportion of patients with anti tumor response to AZD4573. response assessment by Cheson (2014) criteria for for NHL, SLL, T-cell lymphoma and Richter syndrome, IWG criteria for CLL (Hallek 2008) and myeloma (Palumbo 2014), AML response criteria for AML (Doner 2010), SWOG (2016) criteria for ALL and MDS and CMML by IWG (Savona 2015) .Response will be evaluated every 4-12 weeks (based on disease type) until progression
Duration of response (DOR) | From time of first dose until disease progression expected to be for up to 12 months
  To assess the duration of anti tumor activity of AZD4573. To assess the progression free survival of AZD4573. response assessment by Cheson (2014) criteria for for NHL, SLL, T-cell lymphoma and Richter syndrome, IWG criteria for CLL (Hallek 2008) and myeloma (Palumbo 2014), AML response criteria for AML (Doner 2010), SWOG (2016) criteria for ALL and MDS and CMML by IWG (Savona 2015) . Response will be evaluated every 4-12 weeks (based on disease type) until progression
Antitumor activity of AZD4573 in patients by assessing overall survival (OS). | From time of first dose until death or study end whatever is earlier expected to be for up to 12 months
  Proportion of patients alive at 12 months post treatment start or other defined timepoints
Minimal Residual Disease (MRD) | From time of first dose until discontinuation of AZD4573 expected to be for up to 12 months
  For applicable histologies/disease indications (e.g., CLL) using IWG criteria for response assessment every 4-12 weeks from start of treatment.
Progression free survival (PFS) | From time of first dose until first observation of progression expected to be for up to 12 months
  To assess the progression free survival of AZD4573. response assessment by Cheson (2014) criteria for for NHL, SLL, T-cell lymphoma and Richter syndrome, IWG criteria for CLL (Hallek 2008) and myeloma (Palumbo 2014), AML response criteria for AML (Doner 2010), SWOG (2016) criteria for ALL and MDS and CMML by IWG (Savona 2015) . Response will be evaluated every 4-12 weeks (based on disease type) until progression

CONTACTS AND LOCATIONS:
Locations (12):
- Germany (5):
  - Research Site, Aachen
  - Research Site, Bonn
  - Research Site, Göttingen
  - Research Site, Heidelberg
  - Research Site, Ulm
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Nieuwegein
- United Kingdom (5):
  - Research Site, Cardiff
  - Research Site, Manchester
  - Research Site, Plymouth
  - Research Site, Southampton
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Cidado J, Boiko S, Proia T, Ferguson D, Criscione SW, San Martin M, Pop-Damkov P, Su N, Roamio Franklin VN, Sekhar Reddy Chilamakuri C, D'Santos CS, Shao W, Saeh JC, Koch R, Weinstock DM, Zinda M, Fawell SE, Drew L. AZD4573 Is a Highly Selective CDK9 Inhibitor That Suppresses MCL-1 and Induces Apoptosis in Hematologic Cancer Cells. Clin Cancer Res. 2020 Feb 15;26(4):922-934. doi: 10.1158/1078-0432.CCR-19-1853. Epub 2019 Nov 7. PMID 31699827